CLINICAL TRIAL: NCT01790750
Title: Pocket Echocardiography System (PES) for Detection of Patent Ductus Arteriosus (PDA) in Neonates
Brief Title: Pocket Echocardiography System (PES) for Detection of PDA in Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: IRB201200340
Record Dates: First submitted 2013-02-11; First posted 2013-02-13 (Estimated); Results first posted 2014-04-11 (Estimated); Last update posted 2014-04-11 (Estimated); Status verified 2014-03

CONDITIONS: Patent Ductus Arteriosus
Keywords: PDA; Echo; PES; Handheld echo system
MeSH Terms: conditions — Ductus Arteriosus, Patent

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PES first, then FFES (Other): A 5-minute Pocket echocardiography system scan (PES) scan will be performed to detect PDA on neonates. This scan will be followed by a Full Featured Echocardiography System Scan (FFES) and scan results will be compared.
  Interventions: Device: PES first, then FFES

INTERVENTIONS:
Device: PES first, then FFES — A 5-minute Pocket echocardiography system scan (PES) scan will be performed to detect PDA on neonates. This scan will be followed by a Full Featured Echocardiography System Scan (FFES) and scan results will be compared.
  Other Names: Pocket echocardiography system scan; Full Featured Echocardiography System Scan

SUMMARY:
This is a single-center, feasibility study involving all neonates admitted to the neonatal intensive care unit with orders for a cardiac echo evaluation. Parents will be approached and provided a description of the study. No written consent will be requested, but parents have the option of opting out. Each patient will have a 5 minute Pocket echocardiography system scan followed by a full echo performed on a traditional full featured echo system. The objective is to assess if the current Food and Drug administration (FDA) approved Pocket echocardiography system (PES) can detect patent ductus arteriosus (PDA) in neonates as comparable to traditional full featured echo systems (FFES) and/or physical exam alone.

DETAILED DESCRIPTION:
All newborns admitted to the neonatal intensive care unit with orders for a cardiac echo evaluation will be included in this study. Parents will be approached and provided a description of the study. No written consent will be requested, but parents have the option of opting out. If parents agree to be part of this study, a 5-minute PES scan will be performed first so as to not bias the sonographer. Then, a full echocardiogram study will be performed on a traditional FFES. The scans will be performed at the bedside. The images will be reviewed and compared by fellow and/or attending and by experienced sonographer. The scans will include short axis view, ductal view and arch view.

The objective of the study is to assess if the current FDA approved PES can detect PDA in neonates as comparable to traditional full featured echo systems and/or physical exam alone. Using PES for PDA diagnosis will be an accessible, economic and effective way of complementing the findings in our physical exam by increasing diagnostic accuracy, and detecting PDA's at the bedside comparable to a full size traditional echocardiographic system.

ELIGIBILITY:
Inclusion Criteria:

* All newborn infants with orders for cardiac echocardiography evaluation in clinically stable condition

Exclusion Criteria:

* Known congenital heart disease.
* Clinically unstable (Meaning by unstable patients: Those patients that need cardiopulmonary resuscitation, or in maximum ventilatory or inotrope support and in immediate need for Extracorporeal Membrane Oxygenation or major surgery or whenever the physician attending responsible for the clinical care of the patient considers that a traditional echo needs to be done urgently)

Ages: 1 Day to 90 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2013-02; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Curt DeGroff, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recruited in the NICU.
Period: Overall Study
Arm/Group | PES First, Then FFES
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | PES First, Then FFES
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 50
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: weeks] | 34.8 (4.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 33
Region of Enrollment [Number; unit: participants]
  United States | 50
Body Weight [Mean (Standard Deviation); unit: kg] — Mean body weight
  kg | 2.470 (1.157)

OUTCOME MEASURES:

1. Primary Outcome: False Positives Results of Pocket Echocardiography System (PES) Detection of Patent Ductus Arteriosus (PDA) to Full Featured Echo System (FFES)
Description: Evaluate the usefulness of the currently FDA approved Pocket Echocardiography System (PES) in PDA detection as compared to Full Featured Echo System (FFES) by looking at false positives between the two systems.
Time Frame: at baseline
Measure: Mean (Standard Deviation); unit: percentage of false positives
Groups:
- PES First, Then FFES: A 5-minutePocket Echocardiography System Scan (PES) scan will be performed to detect PDA on neonates. This scan will be followed by a Full Featured Echocardiography System Scan (FFES) and scan results will be compared.
Arm/Group | PES First, Then FFES
Number analyzed (Participants) | 50
percentage of false positives | 10.8 (1.2)

2. Primary Outcome: False Negative Results of Pocket Echocardiography System (PES) Detection of Patent Ductus Arteriosus (PDA) to Full Featured Echo System (FFES)
Description: Evaluate the usefulness of the currently FDA approved Pocket Echocardiography System (PES) in PDA detection as compared to Full Featured Echo System (FFES) by looking at false negatives between the two systems.
Time Frame: at baseline
Measure: Mean (Standard Deviation); unit: percentage of false negative
Arm/Group | PES First, Then FFES
Number analyzed (Participants) | 50
percentage of false negative | 3.75 (4.63)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for 3 months.
Arm/Group | PES First, Then FFES
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes